CLINICAL TRIAL: NCT04898647
Title: Clinical Study of the Hyperviscosity Syndrome in Waldenström Macroglobulinemia
Acronym: SLPRaresHvisc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Saint Vincent (Unknown); Centre Henri Becquerel (Other); University Hospital, Caen (Other); University Hospital, Lille (Other); Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0109
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hyperviscosity Syndrome; Waldenstrom Macroglobulinemia
Keywords: Hyperviscosity Syndrome; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with confirmed HVS (Experimental): presence of unexplained elsewhere fundoscopic abnormalities AND either IgM concentration above 30 g/L (densitometry) or cryoglobulin activity
  Interventions: Other: fundoscopic picture; Biological: blood sample; Procedure: bone marrow sample
- Patients with confirmed absence of HVS (Active Comparator)
  Interventions: Other: fundoscopic picture; Biological: blood sample; Procedure: bone marrow sample
- Remaining patients (Experimental)
  Interventions: Other: fundoscopic picture; Biological: blood sample; Procedure: bone marrow sample

INTERVENTIONS:
Other: fundoscopic picture — A central review of numerised fundoscopic picture will be performed.
Biological: blood sample — Two 10 ml blood vials will be sampled in addition to standard blood sampling for getting 6 to 7 200 μL aliquot.
  One 5 ml EDTA vial for GP1bα expression study, only if this sample can be sent to hemostasis laboratory within the 4 hours after sampling
Procedure: bone marrow sample — Five to 10 ml bone marrow sample will be collected in addition to standard bone marrow sampling for getting molecular characteristics of WM

SUMMARY:
Walsdenström Macroglobulinemia (WM) is defined by a bone marrow lymphoplasmacytic infiltration and the presence of a monoclonal immunoglobulin M (IgM) in blood. Clinical manifestations of the hyperviscosity syndrome (HVS) are related to the large amount of IgM in circulating blood or to some physicochemical characteristics such as the presence of a cryoglobulin property. Although HVS is one of the most frequent criteria for initiating therapy in WM, few studies focused on its description and no diagnostic criteria are available.

The present study aims to identify a diagnostic system for HVS, taking into account objective symptoms such as bleedings, fundoscopic findings and also subjective symptoms such as fatigue and comorbidities that may influence the severity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with WM
* Patients that may require a first-line or subsequent-line therapy
* patients who will require treatment initiation
* patients with serum monoclonal component concentration greater than 15 g/L and who will underwent hyperviscosity assessment, even if hyperviscosity is not found and in the absence of other treatment criteria, no treatment is finally initiated.
* Patients agreeing to give informed consent.

Exclusion Criteria:

* Patients with another chronic B-cell malignancy
* patients with lymphoplasmacytic proliferations
* patients with marginal zone lymphoma.
* patients with WM and histologic transformation
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between items collected in questionnaires and HVS detection | 3 years
  Correlation between items collected in questionnaires and HVS detection. Questionnaires are An oncogeriatric form for geriatric assessment, a comorbidity assessment form, a fatigue and quality of live assessment form, and an hemorrhagic assessment form.
Correlation between fundoscopic findings and HVS detection | 3 years
  Correlation between fundoscopic findings and HVS detection

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No